CLINICAL TRIAL: NCT04520334
Title: A Zhineng Qigong Intervention for Patients With Chronic Low Back Pain and/or Leg Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: The Swedish Institute for Health Sciences (Unknown); Ekhaga foundation (Unknown); Greta and Johan Kock Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Project Zhineng Qigong
Record Dates: First submitted 2014-03-03; First posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Chronic Low Back Pain; Chronic Sciatica; Lumbar Spinal Stenosis; Lumbar Disc Herniation; Lumbar Spondylolisthesis; Lumbago; Lumbar Disc Degeneration; Persistent Postoperative Pain
Keywords: Exercise; Training; Qigong; Clinical Trial
MeSH Terms: conditions — Spinal Stenosis; Intervertebral Disc Displacement; Spondylolisthesis; Low Back Pain; Intervertebral Disc Degeneration; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Zhineng Qigong (Other): Zhineng Qigong intervention
  Interventions: Other: Zhineng Qigong intervention

INTERVENTIONS:
Other: Zhineng Qigong intervention — The intervention consisted of group activities which were performed in one group, as lectures, demonstrations, and Zhineng Qigong training, all planned and led by European Zhineng Qigong.
  The group activities were performed during four weekends (12 hours each) and weekly training two times per week (each for two hours). Introductory lecture (two hours) was given at the evening before the first weekend. The respondents were recommended daily Zhineng Qigong training with help of an instructional training CD.

SUMMARY:
The purpose of this study is to evaluate a Zhineng Qigong intervention for patients with chronic low back pain and/or leg pain, and to test feasibility aspects.

DETAILED DESCRIPTION:
Zhineng Qigong is a self-training method which enables the participant to take an active part in a possible recovery process.

The aims of this study are: 1) evaluate a Zhineng Qigong intervention regarding health aspects (both subjective and objective outcomes) in patients with chronic low back pain and/or leg pain; 2) test different aspects of feasibility including recruiting from different patient populations and testing outcome measurements; and, 3) get a basis for power calculation for a future Randomised Controlled Trial.

Based on previous experiences after Zhineng Qigong training with European Zhineng Qigong, this study is based on the following hypotheses:

1. Zhineng Qigong training gives pain reduction and reduced consumption of analgesics.
2. Zhineng Qigong training reduces lumbar spine-related symptoms (other than pain).
3. Zhineng Qigong training reduces healthcare utilisation, including lumbar spine surgery.
4. Zhineng Qigong training improves walking ability, mobility, and functional capacity.
5. Zhineng Qigong training improves Health-Related Quality of Life, including perceived concentration ability, distress, sleeping quality, vitality, depression, mood, and anxiety.

The investigators´ idea was to give patients with chronic low back pain and/or leg pain the opportunity to practise Zhineng Qigong in an intervention arranged by European Zhineng Qigong. To this prospective interventional study without control group, patients were recruited from the Swedish spine surgery register (SweSpine), Orthopaedic clinic, and Primary Healthcare. The intervention period was 12 weeks, with measurements once before and once after intervention. However, because of difficulties in recruiting, 15 of the respondents were enrolled to 3 weeks shorter intervention, joining respondents who already started the 12 weeks intervention. Totally, 55 respondents were enrolled.

Background data:

* Age
* Gender
* Marital status
* Children at home (number and age)
* Duration of symptoms in the lumbar spine and/or leg (year-month when the symptoms started)
* Lumbar spine diagnosis (name and year-month of the diagnosis)
* History of lumbar spine surgery (number of times and which years)
* Type of surgery and surgery level(s) (for postoperative patients)
* Sick- or disability pension (since which year-month and main reason)
* Treatments and/or training methods already tried (also for how long time)
* Educational level
* Occupation or living situation
* Smoking habits
* Financial difficulties

The same physiotherapist examined the respondents once before and once after the intervention period. Two weeks before and two weeks after the intervention period, a "pain diary" was filled in by the respondents. Also, they filled in questionnaires once before and once after the intervention.

During the intervention period participation in the group activities was registered on an attendance list. Every day during the intervention period and two weeks after, the respondents filled in a "training diary" with information about how much Zhineng Qigong was practised besides the group activities.

The respondents that were on waiting list for lumbar spine surgery were asked by telephone if lumbar spine surgery was performed or not. This was done six months after the intervention was completed.

Descriptive and analytical statistics are used to present the results.

ELIGIBILITY:
General inclusion criteria:

* Low back pain and/or leg pain (caused by lumbar disorder) with at least 3 months duration.
* Pain intensity in lumbar spine and/or leg (caused by lumbar disorder) at least 30 on a 0-100 Visual Analogue Scale (VAS), being "the best description of pain the past 2 weeks". (As enrolment initially went slow, also patients scoring VAS pain intensity 25 to 30 became eligible if their pain situations were qualitatively assessed severe, resulting in enrolment of 5 such patients).
* Resident in the county of Skåne (southern part of Sweden).
* Comfortable with the Swedish language.
* Acceptance not to practise Yoga, Meditation, or any other Qigong exercises during or 1 month after the intervention.

Specific inclusion criteria, clinical pathway:

* Postoperative after lumbar spine surgery: one lumbar spine surgery 1-6 years earlier, for either spinal stenosis, spondylolisthesis, or segmental pain. Pain intensity (back and/or leg) at least 30 on 0-100 mm VAS in latest SweSpine follow-up protocol.
* Patients from Primary Healthcare Centres: chronic low back pain (at least 3 months duration) with or without leg pain.
* Patients on waiting list for lumbar spine surgery: Planned first surgery for either spinal stenosis, spondylolisthesis, or segmental pain.

Exclusion criteria:

* Lumbar spine or other major surgery planned before, during, or within 1 month after the intervention period.
* History of serious mental disease, epilepsy, or narcolepsy.
* Current abuse of medicament, drug, or alcohol.
* Pregnancy (due to practical reasons only).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Filled in once daily during 2 weeks, directly before and directly after the intervention period, respectively
  "Pain diary" (designed for this study) measured most usual pain intensity (NRS; 0-10) in lumbar spine and/or leg (caused by lumbar spine disorder).

SECONDARY OUTCOMES:
Pain symptoms | Before intervention and as soon as possible after
  Question (designed for this study) with checkboxes for selecting common lumbar spine-related pain symptoms.
Non-pain symptoms | Before intervention and as soon as possible after
  Question (designed for this study) with checkboxes for selecting common lumbar spine-related non-pain symptoms.
How often "free from pain" | Before intervention and as soon as possible after
  Question (designed for this study) with options "Almost never" to "Completely free".
How often "free from non-pain symptoms" | Before intervention and as soon as possible after
  Question (designed for this study) with options "Almost never" to "Completely free".
Change in intake of analgesics | At baseline concerning past 3 months, after intervention since intervention start
  Question (designed for this study) with options.
Change in intake of other medications | At baseline concerning past 3 months, after intervention since intervention start
  Question (designed for this study) with options.
Healthcare utilisation | At baseline concerning past 3 months, after intervention since intervention start
  Number of visits to physicians, nurses, physiotherapists, occupational therapists, and others. Question designed for this study.
Performed lumbar spine surgery | 6 months after intervention
  Follow-up if planned surgery was performed, for respondents on waiting list for lumbar spine surgery.
Walking ability | Before and after the intervention period
  The respondent walked 10 meters and back, gait performance was noted ("normal gait", "slight limping", or "severe limping").
Active cervical range of motion | Before and after the intervention period
  Flexion, extension, rotation, and lateral flexion measured using Myrin inclinometer.
Active maximal functional shoulder mobility | Before and after the intervention period
  Active shoulder flexion and "hand on neck" were measured using goniometer. "Hand on back" position was noted ("buttocks"; "lumbosacral"; "thoracolumbar"; and, "between scapulae").
Passive hip mobility | Before and after the intervention period
  Hip flexion, and external and internal rotation were measured using goniometer. Extension was assessed as normal or reduced.
Finger tip-floor distance | Before and after the intervention period
  Flexion of lumbar spine with straight knees, with direction of fingers towards the floor in front of the feet. The distance between the middle finger tips and the floor was measured using tape measure.
Schober test | Before and after the intervention period
  The respondent was asked to do a lumbar flexion with straight knees to a self-chosen range and the increased distance between two skin marks (made at level S1 and 10 centimetres cranially) was registered using tape measure.
Single leg stance | Before and after the intervention period
  A functional test for balance. The respondent lifted each foot to a standard height of 20 centimetres and tried to maintain the position for 30 seconds. Timed scores were recorded with a digital stop watch.
Timed get-up-and-go | Before and after the intervention period
  A test for functional mobility. The respondent sat in a chair and at a verbal signal, the respondent stood up without using hands and walked to a point 3 meters in front, then turned around, walked back and sat down again without using hands. Timed scores were recorded with a digital stop watch.
Straight leg raising test | Before and after the intervention period
  The flexion angle of each hip was measured using Myrin inclinometer placed on the ankle joint. Also, eventual pain radiating to the leg and/or low back pain was registered.
Oswestry Disability Index version 2.1a | Before intervention and as soon as possible after
  Questionnaire assessing spine-related disability "for today".
Short Form 36 version 2 | Before intervention and as soon as possible after
  Questionnaire assessing generic Health-Related Qualify of Life (standard 4-week recall).
EQ-5D-5L (including EQ VAS) | Before intervention and as soon as possible after
  Questionnaire assessing generic Health-Related Qualify of Life "for the day".
Additional aspects concerning Health-Related Qualify of Life | Before intervention and as soon as possible after
  Questions (designed for this study) evaluating perceived concentration ability, distress, sleeping quality, energy level, sadness/depression, irritability, and tension/anxiety, respectively, "the past week" (NRS; 0-10).
Recruitment rate | Before intervention
  The percentage of enrolled patients among those who early were estimated to be eligible.
Retention rate | After intervention
  The percentage of patients who completed the study among those who were enrolled.
Attendance in group activities | During intervention
  Attended hours in group activities were registered.
Individual Zhineng Qigong training time | During intervention and 2 weeks after intervention
  Training diary (designed for this study) with individual daily Zhineng Qigong training time (minutes), besides group activities.
Ability to collect outcome measures | At baseline and after intervention
  The percentage of completed outcome measures.

OTHER OUTCOMES:
Concomitant disorders | Before intervention and as soon as possible after
  Concomitant disorders/major health complaints/symptoms other than related to the lumbar spine. Question designed for this study, with checkboxes for common disorders.
Physical activities | At baseline concerning past 3 months, after intervention since intervention start
  Type and amount of performed physical activities, question designed for this study.
Treatments | At baseline concerning past 3 months, after intervention since intervention start
  Type and amount of received treatments, question designed for this study.
Work status | Before intervention and as soon as possible after
  Work status (Full-time, Part-time, Not working), and the reason not to work full-time. Question designed for this study.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella Pozarek, MD, Principal Investigator — Faculty of Medicine, Department of Health Sciences, Lund University, Sweden
Locations (9):
- Sweden (9):
  - Primary Healthcare Centre Dalby, Dalby
  - Primary Healthcare Centre Löddeköpinge, Löddeköpinge
  - Primary Healthcare Centre Capio Citykliniken Clemenstorget, Lund
  - Primary Healthcare Centre Laurentiikliniken, Lund
  - Primary Healthcare Centre Linero/Östra Torn, Lund
  - Primary Healthcare Centre Måsen, Lund
  - Primary Healthcare Centre Nöbbelöv, Lund
  - Orthopaedic clinic, Skåne University Hospital, Malmo
  - Primary Healthcare Centre Södra Sandby, Södra Sandby

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pozarek G, Stromqvist B, Ekvall Hansson E, Ahlstrom G. Pain and function in patients with chronic low back pain and leg pain after Zhineng Qigong - a quasi-experimental feasibility study. BMC Musculoskelet Disord. 2023 Jun 13;24(1):480. doi: 10.1186/s12891-023-06581-w. PMID 37312140